CLINICAL TRIAL: NCT02539251
Title: Adaptation and Validation of the Ages and Stages Questionnaires -3 (ASQ-3) in Arabic
Brief Title: Arabic Ages and Stages Questionnaire-III
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Lama Charafeddine, Assistant Professor of Clinical Pediatrics Fellowship Program, MD FAAP, American University of Beirut Medical Center
Other Study IDs: PED.LC.07
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Child Development
Keywords: Early Child Development; Ages and Stages Questionnaire _3; Validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Validation of Arabic ASQ-3: This group of patients will serve as a reference for validation of the Arabic ASQ-3
  Interventions: Behavioral: Arabic ASQ -3

INTERVENTIONS:
Behavioral: Arabic ASQ -3 — Administration of a developmental questionnaire in Arabic (A-ASQ-3) and validation using BSID-III as a gold standard

SUMMARY:
Early detection and intervention for developmental delays are crucial in promoting healthy child development, hence the need for formal screening. In the Arabic speaking population developmental screening tools are scarce in the native language and there is a need for such a tool for pediatricians and health care workers to use routinely.

This study aims to translate, adapt and validate the newest version of ASQ (ASQ-3) to Arabic (A-ASQ-3) based on the previously published study showing that ASQ-2 was culturally sensitive.

The previously translated A-ASQ-2 will be revised and updated to match the new ASQ-3, then revised by experts in child development. Questionnaires will be adapted and field-tested on 15 subjects per age group (total of 75). For validity, the revised version will be tested on 500 Lebanese children (100 children per age group) selected from all Lebanese governates.

It is expected to generate a culturally adapted and validated Arabic tool for screening children for any developmental delay up to 3 years of age. This tool once published will be available for use by primary care providers and caregivers in Arabic speaking countries. It may be used to screen children for developmental delay as early as 7 months therefore prompting prevention of further delay by starting early intervention and promoting child development.

DETAILED DESCRIPTION:
The Ages and Stages Questionnaires (ASQ) is a developmental screening questionnaire for parents to answer regarding their children's level of growth and development between the ages of 7 months and 3 years. This questionnaire was translated into Arabic in order to adapt it for the Arab speaking culture. For the first phase of this study, aiming to adapt and field-test this translated version, parents of eligible children will be recruited from the AUBMC outpatient clinics (OPD and Private Clinics). Interested parents of eligible children will be invited to a private meeting in private settings where the study will be thoroughly explained. 75 parents (fathers or mothers) will be interviewed and asked to answer the ASQ.

At a later stage, 500 parents will be interviewed and asked to answer the ASQ in order to test its validity. A list of all day care centers in Lebanon will be retrieved from the ministry of public health website and a list of all Lebanese pediatricians will be sought from the both Lebanese Order of Physicians (Beirut and Tripoli). Eligible day cares are the ones with at least 15 children between 7 and 36 months. Eligible physicians are those who are actively seeing patients aged between 7 and 36 months with a patient load of at least 10 per day.

To minimize selection bias and to include different socioeconomic groups, a random sample of eligible day care centers and pediatricians from across the Lebanese governorates (Beirut, Mount Lebanon, South Lebanon, North Lebanon and Beqaa) will be selected.

After obtaining the permission of the selected day care centers and pediatricians, flyers explaining the study and inviting parents to participate will be distributed and posted at those centers. Parents of eligible children who contact us and show interest in participating will be invited for a meeting in private settings. Construct validation will be done using varimax rotation, concurrent validity will be done by correlating ASQ-3 scores with Bayley scale for infant development scores. Sensitivity and specificity will also be tested.

Parents will be asked some questions regarding their child's growth in order to evaluate several aspects of his/her developmental skills. It takes 10-15 minutes to complete the questionnaires. After completing the questionnaire, the child's developmental status will be evaluated and any risk of delay will be detected.

ELIGIBILITY:
Inclusion Criteria:

Adaptation:

* Arabic speaking parents of children between the ages of 4 months and 3 years

Validation:

* Children between 4 months and 3 years of age in chosen day care centers
* Children between 4 months and 3 years of age presenting to their pediatricians offices for well child check up.

Exclusion Criteria:

* Children with known severe disability
* Children with chronic condition that might interfere with the developmental testing (blindness, deafness, congenital hypothyroidism, severe mental disability)

Ages: 4 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For adaptation, 75 parents of eligible children between the ages of 4 months and 3 years will be approached.
  For validation of A-ASQ-3, 500 Children (100 per age group) from a random sample of day care centers and pediatricians' clinics from across the country will be recruited.
Sampling Method: Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Adapt and validate Arabic ASQ by measuring construct validity (varimax rotation), concurrent validity by correlating ASQ-3 scores with BSID-III scores and computing sensitivity and specificity taking BSID-III as gold standard. | 2 years
  After cultural adaptation, Arabic ASQ-3 will be validated by measuring construct validity using varimax rotation, concurrent validity by correlating ASQ-3 scores with Bayley scale for infant development scores and by computing the Arabic ASQ-3 sensitivity and specificity taking BSID-III as gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD FAAP, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Background] Council on Children With Disabilities; Section on Developmental Behavioral Pediatrics; Bright Futures Steering Committee; Medical Home Initiatives for Children With Special Needs Project Advisory Committee. Identifying infants and young children with developmental disorders in the medical home: an algorithm for developmental surveillance and screening. Pediatrics. 2006 Jul;118(1):405-20. doi: 10.1542/peds.2006-1231. PMID 16818591
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735